CLINICAL TRIAL: NCT01294371
Title: Prospective, Multi-Center, Observational Program to Assess Routine Use of Add-back Therapy in Patients With Endometriosis in Russian Federation, Planned for 6-month Course of Gonadoliberin Agonist Lucrin Depot.
Brief Title: Observational Program to Assess Routine Use of Add-back Therapy in Patients With Endometriosis in Russian Federation, Planned for 6-month Course of Lucrin Depot® (Leuprorelin)
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Almedis (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-762
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Results first posted 2013-07-22 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-05

CONDITIONS: Genital Endometriosis
Keywords: Lucrin Depot; genital endometriosis; 6 months therapy

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Leuprorelin: Patients with genital endometriosis received leuprorelin (Lucrin Depot®) in accordance with the respective marketing authorization/manufacturer's directions. All participants received leuprorelin for up to 6 months intramuscularly at a dose of 3.75 mg once a month. If intramuscular administration was not possible, leuprorelin was injected subcutaneously at a dose of 3.75 mg once a month. The first injection was to be carried out on the 3rd day of a menstrual period.
  Accepted options for add-back therapy included: monophasic combined low-dose products for hormonal replacement therapy; combined oral contraceptives; and, if use of hormones was not possible, phytoestrogens with calcium products.

SUMMARY:
The purpose of this study is to assess rates of administration of add-back therapy in patients with endometriosis in the Russian Federation, during a 6-month course of gonadoliberin agonist leuprorelin 3.75 mg.

DETAILED DESCRIPTION:
This was a non-interventional, observational program in which Lucrin Depot (leuprorelin acetate) and add-back therapy (hormone and non-hormone) were prescribed in the usual manner in accordance with the terms of the local marketing authorization with regards to dose, population and indication (for leuprorelin acetate) and with regards to the local guidelines or therapeutic recommendation (for add-back therapy).

The rationale for the study was the necessity to characterize the patient population and long-term leuprorelin acetate administration in the Russian Federation. Further, it was important to characterize the compliance, tolerability, and safety profile of this therapy in the routine clinical care setting in the Russian Federation.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 50 years
* Written Patient Consent for Use/Disclosure of Data
* Diagnosis of genital endometriosis confirmed by laparoscopy (external genital endometriosis) or ultrasound (internal genital endometriosis)
* Candidate for treatment with Lucrin Depot for 6-month course
* Patients with suspected endometriosis suffering from chronic pelvic pain if other reasons for pain are excluded

Exclusion Criteria:

* Contraindications to administration of Lucrin Depot (leuprorelin):

  * Hypersensitivity to leuprorelin similar products of protein origin or any of the excipients in drug product composition
  * Vaginal bleedings of unknown etiology
  * Hysterectomy
  * Pregnancy and lactation
* Menopause (absence of cyclic menstrual hemorrhages for 1 year before the start of this program)
* Acute infectious period, inclusive of acute inflammatory diseases of small pelvic organs
* Other contraindications that make the patients participation impossible (by investigator judgment)
* Previous enrollment in the present program
* Extra-genital endometriosis

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 391 (Actual)
Dates: Start 2011-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Strugovshchikov, MD, Study Director — AbbVie
Locations (28):
- Russia (28):
  - Site Reference ID/Investigator# 51643, Chelyabinsk
  - Site Reference ID/Investigator# 50577, Irkutsk
  - Site Reference ID/Investigator# 50561, Izhevsk
  - Site Reference ID/Investigator# 50560, Kazan'
  - Site Reference ID/Investigator# 50570, Moscow
  - Site Reference ID/Investigator# 50567, Moscow
  - Site Reference ID/Investigator# 50565, Moscow
  - Site Reference ID/Investigator# 50564, Moscow
  - Site Reference ID/Investigator# 62184, Nizhny Novgorod
  - Site Reference ID/Investigator# 50558, Nizhny Novgorod
  - Site Reference ID/Investigator# 50557, Orenburg
  - Site Reference ID/Investigator# 50545, Perm
  - Site Reference ID/Investigator# 53156, Perm
  - Site Reference ID/Investigator# 50547, Saint Petersburg
  - Site Reference ID/Investigator# 50548, Saint Petersburg
  - Site Reference ID/Investigator# 50549, Saint Petersburg
  - Site Reference ID/Investigator# 50551, Saint Petersburg
  - Site Reference ID/Investigator# 50552, Saint Petersburg
  - Site Reference ID/Investigator# 50556, Samara
  - Site Reference ID/Investigator# 50555, Saratov
  - Site Reference ID/Investigator# 50554, Stavropol
  - Site Reference ID/Investigator# 50580, Stavropol
  - Site Reference ID/Investigator# 50579, Tyumen
  - Site Reference ID/Investigator# 50575, Vladivostok
  - Site Reference ID/Investigator# 50562, Volzhskiy, Volgograd Region
  - Site Reference ID/Investigator# 48866, Voronezh
  - Site Reference ID/Investigator# 54502, Voronezh
  - Site Reference ID/Investigator# 50563, Yekaterinburg

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Leuprorelin
Started | 391
Treated | 390
Completed | 357
Not Completed | 34
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 12
Not completed — Lost to Follow-up | 6
Not completed — Administrative Reason | 1
Not completed — Other | 14

BASELINE CHARACTERISTICS:
Arm/Group | Leuprorelin
Number analyzed (Participants) | 391
Age Continuous [Mean (Standard Deviation); unit: years] | 33.8 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 391
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 386
  Asian | 5
Region of Enrollment [Number; unit: participants]
  Russian Federation | 391
Endometriosis location [Number; unit: participants] — Endometriosis is divided into genital and extra-genital by location. Genital endometriosis is internal endometriosis - adenomyosis (endometriosis of the uterus). Extra-genital endometriosis is external endometriosis (endometriosis of the uterine cervix, vagina, retro cervix area, ovaries, fallopian tubes, peritoneum, rectouterine space).
  participants
    External endometriosis | 179
    Internal endometriosis | 108
    Combined type | 104
Time from endometriosis diagnosis [Mean (Standard Deviation); unit: months] | 3.8 (16.7)
Severity of Endometriosis [Number; unit: participants] — Surgically, endometriosis can be staged I-IV (Revised Classification of the American Society of Reproductive Medicine) per the following:
  Stage I (Minimal): Findings restricted to only superficial lesions and possibly a few filmy adhesions;
  Stage II (Mild): In addition, some deep lesions are present in the cul-de-sac;
  Stage III (Moderate): As above, plus presence of endometriomas on the ovary and more adhesions;
  Stage IV (Severe): As above, plus large endometriomas, extensive adhesions.
  participants
    Minimal | 22
    Mild | 74
    Moderate | 180
    Severe | 115

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Administered Add-back Therapy During a 6-month Course of Leuprorelin Treatment
Description: The percentage of participants who received hormone add-back therapy or non-hormone add-back therapy to reduce estrogen deficiency symptom, following local guidelines or therapeutic recommendations, during the 6-month treatment period with leuprorelin.
Time Frame: 6 months
Population: Full Analysis Set included all all patients who had signed the personal authorization form and who administered at least one dose of leuprorelin and who had attended at least one post-baseline visit.
Measure: Number; unit: percentage of participants
Arm/Group | Leuprorelin
Number analyzed (Participants) | 387
percentage of participants
  Any Add-back Therapy Usage | 46.5
  Any Hormonal Add-back Therapy Usage | 21.7
  Any Non-hormonal Add-back Therapy Usage | 26.9

2. Secondary Outcome: Percent Compliance to Treatment With Leuprorelin
Description: Compliance to treatment was calculated as the number of leuprorelin doses administered / number of doses prescribed * 100.
Time Frame: 6 months
Population: Participants who received at least one dose of leuprorelin.
Measure: Mean (Standard Deviation); unit: percent compliance
Arm/Group | Leuprorelin
Number analyzed (Participants) | 390
percent compliance | 96.15 (13.81)

3. Secondary Outcome: Participants With Estrogen Deficiency Symptoms
Description: Estrogen deficiency symptoms include:
  * hot flashes,
  * headaches,
  * palpitations at rest,
  * insomnia,
  * fluctuation of mood.
Time Frame: 6 months
Population: Full Analysis Set
Measure: Number; unit: participants
Groups:
- Overall: Participants with genital endometriosis received leuprorelin in accordance with the respective Marketing Authorization/ Manufacturer's directions for up to 6 months intramuscularly at a dose of 3.75 mg once a month. If intramuscular administration was not possible, leuprorelin was injected subcutaneously at a dose of 3.75 mg once a month. The first injection was carried out on the 3rd day of a menstrual period.
  Accepted options for add-back therapy included: monophasic combined low-dose products for hormonal replacement therapy; combined oral contraceptives; and, if use of hormones was impossible - phytoestrogens with calcium products.
- Plus Add-Back Therapy: Participants with genital endometriosis received leuprorelin in accordance with the respective Marketing Authorization/ Manufacturer's directions, and add-back therapy following local guidelines or therapeutic recommendations.
- No Add-Back Therapy: Participants with genital endometriosis received leuprorelin in accordance with the respective Marketing Authorization/ Manufacturer's directions, and no add-back therapy.
Arm/Group | Overall | Plus Add-Back Therapy | No Add-Back Therapy
Number analyzed (Participants) | 387 | 178 | 209
participants
  Hot Flashes | 303 | 173 | 130
  Headaches | 139 | 94 | 45
  Palpitations at Rest | 100 | 73 | 27
  Overall Insomnia | 190 | 116 | 74
  Fluctuation of Mood | 203 | 113 | 90

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Leuprorelin
Serious Adverse Events (participants affected / at risk) | 0/390
Other Adverse Events (participants affected / at risk) | 0/390

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.